CLINICAL TRIAL: NCT06368531
Title: Long-term Monitoring of Sleep with Ear-EEG in Patients with Chronic Pain
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: T&W Engineering A/S (Industry); University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 2314270
Record Dates: First submitted 2024-03-26; First posted 2024-04-16 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain; Insomnia
MeSH Terms: conditions — Chronic Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Insomnia is reported by more than 50% of patients with chronic pain. In this study, the investigators aim to advance the understanding of physiological sleep in individuals with chronic pain. To do this the investigators will monitor at-home sleep with an ear-EEG over 20 nights in patients with chronic pain and collect self-reported measures of sleep and pain. The collected data will be used to explore and characterize intra-individual variations in sleep metrics (e.g. total sleep time, time in each sleep stage (N1, N2, N3, REM), sleep latency, REM stage latency, wake after sleep onset, sleep efficiency, number of arousals and arousal index) over 20 nights.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible, all inclusion criteria must be answered "yes":

* Understand and write Danish.
* Pain present on most days or every day during the past 3 months.
* Pain limits daily activities or work on some days, most days or every day during the past 3 months.
* Pain intensity equal to or larger than 4 on 0-10 Numeric Rating Scale [NRS] within the last week.
* Informed consent obtained before any study related activities.

Exclusion Criteria:

For a subject to be eligible, all exclusion criteria must be answered "no":

* Previous stroke or cerebral haemorrhage and any other structural cerebral disease.
* Obstructive sleep apnoea (Defined as yes to 3 or more questions in the STOP-BANG questionnaire for women and 4 or more questions for men).
* Teeth grinding (bruxism).
* Pregnancy or lactation (Pregnancy is screened for through self-reporting as no risks regarding pregnancy have been identified for the described study procedures).
* Narrow or malformed ear canals or piercings, making ear-EEG infeasible.
* Allergic contact dermatitis caused by metals or generally prone to skin irritation.
* People judged incapable, by the investigator, of understanding the participant instruction or who are not capable of carrying through the investigation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for this study are individuals with chronic pain in compliance with the inclusion/exclusion criteria listed below. The health status of the subjects is assessed by self-reports.
  Inclusion and exclusion criteria ensure generalizability of study results for a broad population of individuals with chronic pain, and only serious concomitant conditions, which could interfere with the study procedures should prevent subjects from entering the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
sleep period time (SPT) from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Qualitative sleep parameters obtained from sleep diary. | Sleep diary is completed 5 mornings every week for 4 weeks
  Sleep diary is completed in the morning
Pain intensity rating | Pain intensity rating is completed 5 mornings every week for 4 weeks
  Average pain intensity during the last day and current pain intensity in the morning will be assessed on an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (worst imaginable pain)
Time from sleep onset until final awakening (TST) from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Sleep efficiency (SE) from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM). SE is the ratio of TST to time in bed / 100%
Sleep onset latency (SOL) from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Wake after sleep onset (WASO) from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
REM sleep latency from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Time from sleep onset until first epoch of REM stage sleep from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Amount of wake and stage N1, N2, N3, and R sleep as a percentage of SPT from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Number of awakenings within TST from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).
Arousal index which is number of arousals per hour from Ear EEG | 5 nights every week for 4 weeks
  Sleep metrics will be derived from the EEG assessments as recommended by the American Academy of Sleep Medicine (AASM).

SECONDARY OUTCOMES:
Ease-of-use and Comfort with ear EEG | Completed every morning after ear EEG first 2 weeks and at end of study
  Three 0-10 questions are used: 1) How did you experience falling asleep with the ear EEG device, 2) How did you experience sleeping with the ear EEG device?, 3) How would you rate your experience of soreness or discomfort in your ears after sleeping with the device? A lower sum score is worse.
Adverse device effects | Baseline, after 2 weeks, after 6 weeks
  Any adverse device effect defined as an adverse effect related to the use of the ear EEG
Polysomnography | Baseline
  Polysomnography (PSG) is used in this study to ensure that the data that comes out of the automatic ear-EEG based sleep scoring matches the clinicians sleep scores based on the PSG. It will enable further development of the existing algorithm for automating the data analysis.

OTHER OUTCOMES:
Sleep quality | Baseline
  Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI), which is developed to provide a reliable, valid and standardized measure of sleep quality. The PSQI consists of 19 items with 15 multiple choice questions and 4 open-ended questions. The 19 items form the basis a global score. The seven components evaluated by the PSQI are: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medications and daytime dysfunction. Each component has a score ranging from 0 to 3 yielding a total score of 21, with higher scores reflecting worse sleep difficulties
Insomnia | Baseline
  Insomnia will be assessed with the Insomnia Severity Index (ISI) which encompasses seven items measuring severity of sleep-onset; sleep maintenance and early morning awakening difficulties; satisfaction with sleep patterns; daily function interference; impairments due to sleep problems; and distress or concerns due to sleep problems. Each item is rated from 0 to 4 (0 = no problem, 4 = severe problem), yielding a total score of 28, with higher scores reflecting worse insomnia
The Graded Chronic Pain Scale Revised | Baseline
  The Graded Chronic Pain Scale Revised (GCPS-R) is a brief, freely available questionnaire that assesses frequency and severity of pain and its impact. The GCPS-R uses 5 items to categorize pain into mild chronic pain, bothersome chronic pain, and high-impact chronic pain
Age | Baseline
Sex | Baseline
Ethnicity | Baseline
Height | Baseline
Weight | Baseline
Level of education | Baseline
Obstructive sleep apnea | Baseline
  Risk for obstructive sleep apnea (OSA) will be evaluated with the snoring history, tired during the day, observed stop of breathing while sleeping, high blood pressure, BMI > 35 kg/m2 (or 30 kg/m2), age > 50 years, neck circumference > 40 cm and male gender) questionnaire (The STOP-BANG). The STOP-BANG questionnaire is a four item forced yes/no questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Henrik B Vægter, PhD, Principal Investigator — University Hospital Odense
Locations (1):
- Pain Center, Department of Anesthesiology and Intensive Care Medicine, University Hospital Odense, Odense, Denmark

IPD SHARING:
Plan to Share IPD: Undecided